CLINICAL TRIAL: NCT05986383
Title: A Prospective, Multi-center Clinical Study on the Safety and Effectiveness of Chinese Precision Hepatectomy Decision Tree
Brief Title: Multi-center Clinical Study on the Decision Tree of Precision Hepatectomy in China Precision Hepatectomy Decision Tree
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: West China Hospital (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); The First Hospital of Jilin University (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); LanZhou University (Other); Southwest Hospital, China (Other); The Affiliated Hospital of Qingdao University (Other); Affiliated Hospital of Qinghai University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shenzhen People's Hospital (Other); Zhongshan Hospital Xiamen University (Other)
Responsible Party: Principal Investigator, Jiahong Dong，MD, Director, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 21408-0-03
Record Dates: First submitted 2023-03-01; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Primary Liver Cancer; Metastatic Liver Cancer; Benign Liver Neoplasms; Hepatic Echinococcosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Echinococcosis, Hepatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Guoup 1: Liver function is Child Pugh A：If ICG-R15<10%, the standardized residual functional liver volume ratio (RRS) ≥ 40%
- Guoup 2: Liver function is Child Pugh A：If ICG-R15 is 10% - 20%, RRS ≥ 60%
- Guoup 3: Liver function is Child Pugh A：If ICG-R15 is 21% - 30%, RRS ≥ 80%
- Guoup 4: Liver function is Child Pugh A：If ICG-R15 is 31%~40%, only minimal hepatectomy with hepatectomy rate less than 5% can be performed
- Guoup 5: Liver function is Child Pugh A：If ICG-R15>40%, only tumor resection is feasible
- Guoup 6: Liver function is Child Pugh B: only tumor resection is allowed

SUMMARY:
Liver failure (PHLF) after hepatectomy is a relatively serious postoperative complication. Previous studies have shown that liver reserve function is related to PHLF. The "Chinese expert consensus decision tree for hepatectomy" implemented recommends different surgical methods according to the liver function of patients and the standardized residual functional liver volume ratio, so as to achieve accurate hepatectomy and prolong the survival of patients. In the retrospective study, it showed the safety and effectiveness of the decision tree under the condition of extended hepatectomy indications, but it lacked prospective research to evaluate. Therefore, this study intends to evaluate the safety and effectiveness of hepatectomy under the guidance of Chinese expert consensus decision tree through prospective research.

DETAILED DESCRIPTION:
Hepatectomy is an effective treatment for primary liver cancer, with excellent efficacy and controllable safety . The incidence of non fatal complications after Hepatectomy is as high as 45%, ranging from less serious events to life-threatening complications, including infection or sepsis, bleeding, leakage or cardiopulmonary events. Liver Function Insufficiency is a serious complication, which is also described as Post hepatectomy Liver failure (PHLF) after Hepatectomy. PHLF has many definitions. Balzan and his colleagues put forward the "50-50 standard" in 2005, that is, on the fifth day after surgery, total bilirubin>50 μ mol/L (2.9 mg/dl) and prothrombin ratio<50% (INR>1.7) are met simultaneously. The Sensitivity and specificity of this standard are 69.6% and 98.5% respectively , which was confirmed as an effective predictor of death after Hepatectomy in 2009 . The "Edinburgh Standard" proposed by Schindl et al. in 2005 is to divide the severity of PHLF according to Hematology examination and clinical observation, which can be divided into none/mild/moderate/severe . Mullen et al. proposed a peak postoperative bilirubin level>120 μ Mol/L), which can predict the death related to Liver failure, with a sensitivity of 93.3% and a specificity of 94.3% . At present, the 2011 definition of the International Research Group on Hepatosurgery (ISGLS) has been widely used as a standard to describe PHLF. According to the international normalized ratio (INR), hyperbilirubin and other test indicators five days after hepatectomy, and in combination with liver function, kidney function, respiratory function, whether special assessment and special clinical treatment are required, the severity of Liver failure in patients with cirrhosis after Hepatectomy is divided into A, B C has three levels . The reported incidence of PHLF varies greatly, ranging from 0.7% to 34% , but recent reports have more commonly described it as between 8% and 12% . PHLF is an important cause of death after Hepatectomy. In a large study, 70% of all patients who died after liver resection met the PHLF criteria, while over 50% of patients had PHLF as the direct cause of death. Moreover, nearly half of hospital deaths caused by PHLF occur within 30 days after surgery. In addition, the management cost of these postoperative complications is high . Although there are already many treatment strategies that can save patients with PHLF, the evidence for these treatment methods is still limited, and only a few conventional methods are available for clinical use.

Many preoperative factors may lead to PHLF. These have been extensively discussed in other studies, including patient factors, disease pathology, intraoperative characteristics, and postoperative course, but the most important factor that may affect the occurrence of PHLF is the condition of the liver. On the one hand, it is the insufficient amount of remaining liver tissue, accompanied by a decrease in liver regeneration ability in patients with cirrhosis. The morphology, structure, and physiological function of regenerated liver cells are incomplete, which can also affect the function of liver cells. At the same time, postoperative liver reperfusion loss can also lead to insufficient liver functional liver cell count. On the other hand, surgery directly leads to damage to the hepatic vascular structure, changes in microcirculation structure, excessive inflammatory response after surgery leading to liver microcirculation disorders, liver hypoperfusion, and further exacerbating liver injury. Therefore, precise assessment of liver reserve function and monitoring of liver microcirculation disorders during the perioperative period are of great significance for selecting reasonable treatment methods, grasping the safe range of liver resection, and reducing the incidence of postoperative liver failure in patients.

Liver reserve function refers to the additional compensatory potential that the liver can mobilize in response to increased physiological load. In the pathological state of liver damage, the liver reserve function needs to meet the Functional requirement of body metabolism, immunity and detoxification, as well as the needs of liver tissue repair and regeneration. The reserve function of the liver mainly depends on the number of functional liver cell populations and the integrity of their organizational structure. For decades, the Child-Pugh score has been an important prognostic tool for patients with chronic liver disease, used to stratify preoperative risk and to some extent remains a guiding factor for clinical decision-making. The MELD score (the "end stage liver disease model") can better predict the prognosis of chronic liver disease. And MELD score is related to the early prediction of incidence rate and mortality after Hepatectomy. Recently, the albumin bilirubin (ALBI) score and its improvement have been proposed as an objective and evidence-based clinical liver function assessment method. It has been proved to be a reliable assessment of liver dysfunction in many studies , and is found to be superior to Child Pugh score in predicting the outcome after Hepatectomy for liver cancer. The remaining liver volume (FLR) is achieved by calculating the proportion of remaining liver tissue in the total liver volume. To avoid PHLF, based on experience, it is recommended that the FLR be at least 20% of the standard total liver volume, as the remaining parenchyma is normal . In addition, Truant et al. found that patients with residual liver volume (RLV=FLR) related to body weight less than 0.5% of their body weight had a significant risk of postoperative liver dysfunction and death. If the liver is damaged through chemotherapy or existing liver diseases (such as cirrhosis), it is necessary to increase FLR by at least 30% and 40%, respectively .

However, although liver volume itself is important, it may not necessarily be related to liver function. There are inherent limitations to liver capacity and Child Pugh score. Compared to simple calculations of residual liver volume (FLR), the evaluation of functional liver residual volume is better. Among the numerous tests to evaluate functional liver capacity, indocyanine green clearance (ICG R15) is the most commonly used test, which can minimize PHLF and mortality after Hepatectomy. In a large single center study, Professor Yamin strictly applied bilirubin based algorithms and stratified them based on ICG clearance rate, not only deciding which patients to undergo resection, but also deciding which type of resection to perform. In a period of 10 years, excellent results have been achieved, with only one patient having an extremely low mortality rate out of over a thousand resection procedures. However, there are some limitations to ICG clearance, especially in patients with perioperative jaundice and patients with impaired hemodynamics. Another aspect that reflects the reserve function of the liver is the integrity of the tissue structure, which directly determines the microcirculation structure of the liver. The complex functions of liver biosynthesis, metabolism, detoxification, and host defense are closely dependent on a sound liver microcirculation. Research has shown that microcirculation disorders are one of the important pathogenesis of chronic liver disease, running through the entire disease development process. Improving liver microcirculation is beneficial for the recovery of liver function and helps to prevent and delay the formation of liver fibrosis and cirrhosis. The Guidelines for the Diagnosis and Treatment of Liver failure (2012 Edition) mentioned that all kinds of chronic liver disease patients have different degrees of liver microcirculation disorders. Due to the increase of blood viscosity and the slowing of blood flow, the blood perfusion and oxygen supply of microcirculation will inevitably be affected. It is difficult for blood to enter and exit the liver, and the nutritional supply to liver cells cannot be guaranteed, leading to further damage to liver cells, resulting in a vicious cycle. The nutrients absorbed by the gastrointestinal tract are difficult to enter the liver, resulting in indigestion; Drugs absorbed in the bloodstream are difficult to enter the liver and come into contact with liver cells, making it difficult to effectively exert drug efficacy; Metabolic waste is difficult to excrete from the liver, becoming toxins that remain in the liver, leading to liver cell damage and accelerating the progression of liver disease. At present, the main observation indicator reflecting liver microcirculation is effective liver blood flow, which is also the "functional liver blood flow" studied in recent years. Effective Hepatic Blood Flow (EHBF) refers to the blood flow of the liver that comes into contact with liver cells and undergoes material exchange and metabolic function. Under the condition of liver cirrhosis, due to changes in liver microcirculation structure and the establishment of collateral circulation, there is arteriovenous shunt inside and outside the liver. The effective blood flow of the liver (functional liver blood flow) is much lower than the total liver blood flow (physical liver blood flow), and the clearance function of the liver also decreases accordingly. The literature reports that using indocyanine green or D-sorbitol as reagents for EHBF determination showed a significant decrease in EHBF in patients with liver cirrhosis compared to normal individuals. Another study showed that EHBF in patients with chronic liver failure was significantly lower than that in patients with decompensated cirrhosis, and EHBF was closely related to the severity of HBV infection in patients with chronic liver failure, which can be used to predict their 90 day mortality rate. Therefore, EHBF is considered to reflect liver reserve function and also a marker of liver ischemia.

In order to improve the safety of liver resection, establishing a safe and effective liver resection decision tree based on existing experience and data has always been a research direction in liver and gallbladder surgery. In order to avoid Liver failure after Hepatectomy, we should carefully consider whether to retain sufficient functional liver volume before operation. However, there is no uniform standard for clinical hepatobiliary Surgeon to evaluate liver reserve function before Hepatectomy. Each center proposes a variety of hepatectomy decision systems based on Scientific theory and the center's practical experience. At present, most of them refer to the Makuuchi standard of University of Tokyo in Japan, the University of Zurich standard in Europe, the consensus decision tree of Chinese experts on hepatectomy, in addition to Hong Kong, Fudan Zhongshan and other standards.

The evaluation of liver reserve function proposed by the above standards refers to the Child Pugh score, ICG15 minute retention rate (R15), or ICG plasma clearance rate (ICGK). However, the Child Pugh score, ICGR15, and ICGK only reflect the number of functional liver cell populations, and the integrity of liver tissue structure is not directly reflected. EHBF may be able to supplement and improve liver reserve function.

To sum up, previous studies have shown that liver reserve function is related to Liver failure (PHLF) after Hepatectomy. The retrospective study of the Chinese expert consensus decision tree for hepatectomy also shows the safety and effectiveness of the decision tree in the case of expanded hepatectomy indications, but there is a lack of forward-looking research to evaluate it. Therefore, this study intends to evaluate the safety and effectiveness of Hepatectomy under the guidance of the consensus decision tree of Chinese experts through prospective research.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, gender unlimited;
2. Primary liver cancer patients who strictly comply with the clinical diagnostic criteria of the "Guidelines for the Diagnosis and Treatment of Primary Liver Cancer" (2019 version) or who have been confirmed by histopathological or cytological examination, or patients with benign liver neoplasms, or metastatic liver cancer;
3. Child-Pugh liver function rating A/B;
4. ECOG PS score 0-2 points;
5. The liver tumor can be resected (the remaining liver vessel structure is complete, the liver volume is sufficient, and conforms to the decision system of safe hepatectomy);
6. If the patient is HBV antigen positive and the HBV DNA is less than 1.0E+04 IU/ml, routine antiviral treatment is required;
7. Patients with portal hypertension can be included, and the severity can refer to endoscopic esophageal varices or splenomegaly and hypersplenism;
8. Use up to 3 antihypertensive drugs to fully control blood pressure (BP), which is defined as BP<=150/90 mm Hg (mmHg) during screening, and there is no change in antihypertensive treatment within 1 week before the first cycle/day;
9. The patient's expected survival period is more than 3 months;
10. No pregnancy or pregnancy plan;
11. No other contraindications for operation;
12. Subjects voluntarily joined the study and signed the informed consent form, with good compliance and cooperation in follow-up.

Exclusion Criteria:

1. Extrahepatic metastasis of primary liver cancer;
2. Diffuse liver cancer;
3. Suffering from vascular liver diseases such as sinus obstruction syndrome, Budd-Chiari syndrome and congenital vascular malformation;
4. Patients with obstructive jaundice or cholestasis;
5. Preoperative bilirubin>50umol/L (2.9 mg/dL);
6. Pregnant women;
7. Have a history of mental illness or abuse of psychotropic substances;
8. Joint HIV infected patients;
9. With other malignant tumors;
10. Floating population and other patients with poor compliance;
11. Clinical trials involving other experimental drugs or devices within four weeks;
12. The researcher believes that it is not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. CNLC stage Ⅰ a~Ⅱ b -- Ⅲ a (see the indications for hepatectomy of primary liver cancer in the 2019 edition of the diagnostic and treatment specifications for primary liver cancer);
     1. CNLC stage Ⅰ a, Ⅰ b and Ⅱ a liver cancer with good liver reserve function
     2. CNLC stage Ⅱ b liver cancer with tumor localized in the same segment or half of the liver on the same side.
     3. The tumor is limited to the half-liver CNLC stage Ⅲ a liver cancer, and the portal vein branch tumor thrombus (Cheng's classification type I/II).
  2. Patients with benign liver neoplasms;
  3. Patients with metastatic liver cancer.
Sampling Method: Non-Probability Sample
Enrollment: 820 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative liver failure rate (50-50 criteria) | postoperative day 3 and postoperative day 5
  The proportion of patients with Liver failure after Hepatectomy in all patients. Using the 50-50 standard.On the 5th day after surgery

SECONDARY OUTCOMES:
Postoperative liver failure rate (ISGLS criteria) | postoperative day 3 and postoperative day 5
  The proportion of patients with Liver failure after Hepatectomy in all patients. Adopting the ISGLS standard.
Value of indocyanine green retention test at 15 min (ICG-R15) | postoperative day 3 and postoperative day 5
Hepatic effective hepatic blood flow (EHBF) | postoperative day 3 and postoperative day 5
Postoperative remanent liver volume (mL) | postoperative day 5
Volume (mL) of blood loss during the operation | the operation day
Operation time (min) | the operation day
Hepatic inflow occlusion time (min) during the operation | the operation day
Postoperative serum albumin level (g/L) | postoperative day 3 and postoperative day 5
Postoperative serum ALT (U/L) | postoperative day 3 and postoperative day 5
Postoperative serum AsT (U/L) | postoperative day 3 and postoperative day 5
Postoperative serum total bilirubin (umol/L) | postoperative day 3 and postoperative day 5
Postoperative prothrombin time (sec) | postoperative day 3 and postoperative day 5
Postoperative INR value | postoperative day 3 and postoperative day 5
Postoperative periphery platelet amount | postoperative day 3 and postoperative day 5
Postoperative fasting plasma glucose (mmol/L) | postoperative day 3 and postoperative day 5
Child-pugh score | postoperative day 3 and postoperative day 5
Total postoperative complication rate | postoperative day 14
Clavien-Dindo grade of postoperative complications | postoperative day 14